CLINICAL TRIAL: NCT06573619
Title: Therapeutic Adherence in Patients With Chronic Diseases
Acronym: GMAS-MCNT
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 6227 - GMAS-MCNT
Record Dates: First submitted 2024-01-02; First posted 2024-08-27 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Chronic Disease
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Validation of questionnaire — Validation of questionnaire

SUMMARY:
Objectives of the study are:

* The validation of the GMAS questionnaire in patients with chronic disease.
* Measurement of the level of therapeutic adherence in patients with chronic illness.
* Measurement of the level of therapeutic adherence in patients with chronic disease undergoing an experimental trial.

DETAILED DESCRIPTION:
The research is multicentre and will be conducted at the Fondazione Policlinico Gemelli IRCCS in Rome as reference centre together with the other participating centres. Patients will be enrolled at the centres involved, either during visits or during their hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Chronically ill;
* Age 18 years or older;
* Willingness to participate in the study;
* Chronic illness diagnosed at least 3 months before the start of the study;
* Reading and signing the informed consent.

Exclusion Criteria:

* Reduced command of the Italian language;
* Subjects suffering from severe psychiatric disorders;
* Serious clinical conditions that do not permit completion of the questionnaire;
* Refusal to sign the informed consent to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic diseases
Sampling Method: Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2024-01-08 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
The validation of the GMAS questionnaire in patients with chronic disease. | 1 year
  The validation of the GMAS questionnaire in patients with chronic disease.

SECONDARY OUTCOMES:
Measurement of the level of therapeutic adherence in patients with chronic illness. Measurement of the level of therapeutic adherence in patients with chronic disease undergoing an experimental trial. | 1 year
  Measurement of the level of therapeutic adherence in patients with chronic illness.
  Measurement of the level of therapeutic adherence in patients with chronic disease undergoing an experimental trial.

CONTACTS AND LOCATIONS:
Overall Officials: Daniele Napolitano, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Daniele Napolitano, Rome, Italy